CLINICAL TRIAL: NCT01664065
Title: An Open-label, Nonrandomised, Phase I Study to Assess the Pharmacokinetics of Ceftaroline After Intravenous Administration of aSingle Dose of Ceftaroline Fosamil (200 mg) to Patients With End-stage Renal Disease Undergoing Haemodialysis When Compared to a Single Dose of Ceftaroline Fosamil (600 mg)
Brief Title: A Study to Assess the Pharmacokinetics of Ceftaroline in End Stage Renal Disease Patients and Matched Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D3720C00012
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Renal Disease
Keywords: Patient Safety; Tolerability; Pharmacokinetics
MeSH Terms: conditions — Kidney Diseases | interventions — Ceftaroline

ARMS (2):
- AZ drug: A (Experimental): 200 mg Ceftaroline fosamil 1h infusion
  Interventions: Drug: 200 mg Ceftaroline fosamil
- AZ drug: B (Experimental): 600 mg Ceftaroline fosamil 1h infusion
  Interventions: Drug: 600 mg Ceftaroline fosamil

INTERVENTIONS:
Drug: 200 mg Ceftaroline fosamil — 1 h infusion
  Arms: AZ drug: A
Drug: 600 mg Ceftaroline fosamil — 1 h infusion
  Arms: AZ drug: B

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of Ceftaroline in a group of patients with renal disease and matching healthy subjects with normal renal function

DETAILED DESCRIPTION:
An Open-label, Nonrandomised, Phase I Study to Assess the Pharmacokinetics of Ceftaroline After Intravenous Administration of aSingle Dose of Ceftaroline Fosamil (200 mg) to Patients with End-stage Renal Disease Undergoing Haemodialysis when Compared to a Single Dose of Ceftaroline Fosamil (600 mg)

ELIGIBILITY:
Inclusion criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Male and female subjects aged 18 to 75 years (inclusive) with suitable veins for cannulation or repeated venipuncture
* Women of childbearing potential must have a negative pregnancy test, be non-lactating, and be using a highly effective form of birth control for 3 months prior to enrollment, during the study, and for 3 months after completion of all study-related proceed
* Have a body mass index (BMI) between 18 and 35 kg/m2 and weigh at between 50 and 110 kg
* Haematocrit level higher than 30% at screening and baseline for each treatment period

Exclusion criteria:

* History or presence of gastrointestinal, hepatic, or any other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the investigator
* Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG that may interfere with the interpretation of QTc interval changes
* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* Receiving any dialysis treatment other than intermittent haemodialysis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Ceftaroline after intravenous infusion of Ceftaroline Fosamil in patients with end-stage renal disease and a matched control population with normal renal function to characterise the clearance of Ceftaroline. | pre-dose, 20, 40, 60, 65, 75, 90 min, 2.25, 3.25 , 4.25, 5.25, 8, 12, 24, 36, 48 h
  Group 1 (patient group/period 1 and 2); Group 2 (control group - healthy). Maximum plasma concentration (Cmax), time to maximum concentration (tmax), area under the plasma concentration-time curve from zero to infinity (AUC), area under the plasma concentration-time curve from zero to time of the last quantifiable concentration (AUC(0-t)), area under the plasma concentration-time curve from zero to 12 hours after the start of the infusion (AUC(0-12)), terminal rate constant (λz), terminal half-life (t1/2λz),dose normalised Cmax, dose-normalised AUC, dose-normalised AUC(0-t), and dose-normalised AUC(0-12)
Pharmacokinetics of Ceftaroline after intravenous infusion of Ceftaroline fosamil in patients with end-stage renal disease and a matched control population with normal renal function to characterise the clearance of Ceftaroline. | pre-dose, 20, 40, 60, 65, 75, 90 min, 2.25, 3.25 , 4.25, 5.25, 8, 12, 24, 36, 48 h
  Group 1 (patient group/period 1 and 2);Group 2 (control group - healthy). Mean residence time (MRT), total body clearance of drug from plasma (CL for ceftaroline fosamil, apparent CL for ceftaroline), volume of distribution based on the terminal phase (Vz for ceftaroline fosamil, apparent Vz for ceftaroline), volume of distribution at steady-state (Vss for ceftaroline fosamil, apparent Vss for ceftaroline)
Pharmacokinetics of Ceftaroline after intravenous infusion of Ceftaroline fosamil in patients with end stage renal diseaseand to characterise the clearance of Ceftaroline. | pre-dose, 20, 40, 60, 65, 75, 90 min, 2.25, 3.25 , 4.25, 5.25, 8, 12, 24, 36, 48 h
  Group 1 (patient group/period 2). Area under the plasma concentration -time curve from 75 min to 5.25 hr after the start of the infusion (AUC(1-5)), amount of drug extracted unchanged into the dialysate (AD) during each 1-hour interval, cumulatively, and overall (AD(1-5)) for the entire haemodialysis session (time: 75 min to 5.25 hr after the start of infusion); percent of dose recovered in dialysate (fD,%) during each 1-hour interval, cumulatively, and overall (fD(1-5),%) for the entire haemodialysis session (time: 75 min to 5.25 hr after the start of infusion), extraction coefficient (E) at each time point during haemodialysis

SECONDARY OUTCOMES:
Safety and tolerability in terms of adverse events, laboratory data, physical examinations, ECG and vital signs. | Screening up to 10 days after discharge from study site.
Pharmacokinetics of Ceftaroline M-1 after intravenous infusion of Ceftaroline fosamil in patients with end-stage renal disease and a matched control population with normal renal function to characterise the clearance of Ceftaroline. | pre-dose, 20, 40, 60, 65, 75, 90 min, 2.25, 3.25 , 4.25, 5.25, 8, 12, 24, 36, 48 h
  Group 1 (patient group/period 1 and 2); Group 2 (control group - healthy). Maximum plasma concentration (Cmax), time to maximum concentration (tmax), area under the plasma concentration-time curve from zero to infinity (AUC), area under the plasma concentration-time curve from zero to time of the last quantifiable concentration (AUC(0-t)), area under the plasma concentration-time curve from zero to 12 hours after the start of the infusion (AUC(0-12)), terminal rate constant (λz), terminal half-life (t1/2λz),dose normalised Cmax, dose-normalised AUC, dose-normalised AUC(0-t), and dose-normalised AUC(0-12)
Pharmacokinetics of Ceftaroline M-1 after intravenous infusion of Ceftaroline fosamil in patients with end stage renal disease and to characterise the clearance of Ceftaroline. | pre-dose, 20, 40, 60, 65, 75, 90 min, 2.25, 3.25 , 4.25, 5.25, 8, 12, 24, 36, 48 h
  Group 1 (patient group/period 2). Area under the plasma concentration -time curve from 75 min to 5.25 hr after the start of the infusion (AUC(1-5)), amount of drug extracted unchanged into the dialysate (AD) during each 1-hour interval, cumulatively, and overall (AD(1-5)) for the entire haemodialysis session (time: 75 min to 5.25 hr after the start of infusion); percent of dose recovered in dialysate (fD,%) during each 1-hour interval, cumulatively, and overall (fD(1-5),%) for the entire haemodialysis session (time: 75 min to 5.25 hr after the start of infusion), extraction coefficient (E) at each time point during haemodialysis
Pharmacokinetics of Ceftaroline fosamil after intravenous infusion of Ceftaroline fosamil in patients with end-stage renal disease and a matched control population with normal renal function to characterise the clearance of Ceftaroline. | pre-dose, 20, 40, 60, 65, 75, 90 min, 2.25, 3.25 , 4.25, 5.25, 8, 12, 24, 36, 48 h
  Group 1 (patient group/period 1 and 2); Group 2 (control group - healthy). Maximum plasma concentration (Cmax), time to maximum concentration (tmax), area under the plasma concentration-time curve from zero to infinity (AUC), area under the plasma concentration-time curve from zero to time of the last quantifiable concentration (AUC(0-t)), area under the plasma concentration-time curve from zero to 12 hours after the start of the infusion (AUC(0-12)), terminal rate constant (λz), terminal half-life (t1/2λz),dose normalised Cmax, dose-normalised AUC, dose-normalised AUC(0-t), and dose-normalised AUC(0-12)
Pharmacokinetics of Ceftaroline fosamil after intravenous infusion of Ceftaroline fosamil in patients with end-stage renal disease and a matched control population with normal renal function to characterise the clearance of Ceftaroline. | pre-dose, 20, 40, 60, 65, 75, 90 min, 2.25, 3.25 , 4.25, 5.25, 8, 12, 24, 36, 48 h
  Group 1 (patient group/period 1 and 2);Group 2 (control group - healthy). Mean residence time (MRT), total body clearance of drug from plasma (CL for ceftaroline fosamil, apparent CL for ceftaroline), volume of distribution based on the terminal phase (Vz for ceftaroline fosamil, apparent Vz for ceftaroline), volume of distribution at steady-state (Vss for ceftaroline fosamil, apparent Vss for ceftaroline).

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, MD, Study Director — AstraZeneca Pharmaceuticals;C2C-716 1800 Concord PikePO. Box 15437Wilmington De 19850-5437; Arpeat Kaviya, MBChB, MRCP, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital 6 Newcomen St; Mirjana Kujacic, MD, Study Chair — AstraZeneca Research and Development SE-431 83 Mölndal
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Background] Sunzel M, Learoyd M, Li J, Li Y, Ngo N, Edeki T. An open-label, non-randomised, phase 1, single-dose study to assess the pharmacokinetics of ceftaroline in patients with end-stage renal disease requiring intermittent haemodialysis. Int J Antimicrob Agents. 2015 Dec;46(6):682-8. doi: 10.1016/j.ijantimicag.2015.09.009. Epub 2015 Oct 22. PMID 26545441
- [Derived] Das S, Li J, Iaconis J, Zhou D, Stone GG, Yan JL, Melnick D. Ceftaroline fosamil doses and breakpoints for Staphylococcus aureus in complicated skin and soft tissue infections. J Antimicrob Chemother. 2019 Feb 1;74(2):425-431. doi: 10.1093/jac/dky439. PMID 30380060
- See also: D3720C00012_SCR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1377&filename=D3720C00012_Study_Synopsis.pdf
- See also: D3720C00012 revised csp REDACTED 13Aug2014 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1377&filename=D3720C00012-revised-csp-1_REDACTED_13_Aug_2014.pdf